CLINICAL TRIAL: NCT06648720
Title: Efficacy and Safety of Shortening Dual Antiplatelet Therapy Duration with IVUS Guidance in PCI Patients: a Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Shortening Dual Antiplatelet Therapy Duration with IVUS Guidance in PCI Patients
Acronym: SHORTDAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Vu Hoang Vu, Head of Interventional Cardiology Department, PhD MD, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHORTDAPT IVUS Trial
Record Dates: First submitted 2024-10-03; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Coronary Arterial Disease (CAD); Percutaneous Coronary Intervention (PCI); Intravascular Ultrasound; Dual Antiplatelet Therapy
Keywords: Shortening DAPT duration; Intravascular Ultrasound (IVUS); Percutaenous Coronary Intervention (PCI); Coronary Arterial Disease (CAD)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (1-Month DAPT): DAPT De-escalation (Intervention Group) (Experimental): Patients in this group will receive DAPT (aspirin and a P2Y12 inhibitor) for 1 month, followed by monotherapy with a P2Y12 inhibitor for the remaining 11 months.
  Interventions: Drug: DAPT de-escalation
- Group 2 (12-Month DAPT): Standard DAPT (Control Group) (No Intervention): Patients in this group will continue with DAPT (aspirin and a P2Y12 inhibitor) for the full 12 months.

INTERVENTIONS:
Drug: DAPT de-escalation — Patients in this group will receive DAPT (aspirin and a P2Y12 inhibitor) for 1 month, followed by monotherapy with a P2Y12 inhibitor for the remaining 11 months.
  Arms: Group 1 (1-Month DAPT): DAPT De-escalation (Intervention Group)

SUMMARY:
This study is designed to assess the efficacy and safety of de-escalating dual antiplatelet therapy (DAPT) at 1 month compared to the standard 12 months of therapy in patients undergoing percutaneous coronary intervention (PCI) guided by intravascular ultrasound (IVUS). The main outcomes measured will include major adverse cardiovascular and cerebrovascular events (NACCE), bleeding events, and target vessel failure (TVF). The goal is to evaluate whether a shorter duration of DAPT is non-inferior to the standard 12-month regimen in preventing ischemic events while reducing the incidence of bleeding.

DETAILED DESCRIPTION:
This multicenter, double-blind, randomized controlled trial will evaluate the clinical outcomes of DAPT de-escalation at 1 month compared to 12 months, in patients who have undergone PCI with drug-eluting stent (DES) implantation. The study aims to optimize post-PCI treatment duration while reducing associated risks such as bleeding complications. Intravascular ultrasound (IVUS) will be used to guide stent placement and optimize results, especially in high-risk, complex cases.

Participants will be randomly assigned to two groups:

1. One month of DAPT, followed by monotherapy with a P2Y12 inhibitor.
2. Standard 12 months of DAPT. Patients will be followed for 12 months after the intervention to track cardiovascular events, bleeding complications, and overall safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients undergoing percutaneous coronary intervention (PCI) with drug-eluting stents (DES).
* Patients with the following clinical indications for PCI:

  * Unstable Angina: Prolonged chest pain at rest, new-onset angina within the past 2 months, or increasing frequency/severity of angina attacks.
  * Acute Myocardial Infarction (MI): With or without ST-elevation.
  * Chronic Coronary Syndrome: Requiring coronary revascularization.
* Patients who agree to participate and provide informed consent.

Exclusion Criteria:

* Inability to Provide Informed Consent: Patients who are unable or unwilling to provide consent.
* Neurological Complications: Stroke or any permanent neurological deficits within the last 3 months.
* Coronary Artery Bypass Graft Surgery: History of CABG surgery.
* Planned Surgery: Patients who have surgeries planned within the next 12 months.
* Severe Chronic Kidney Disease: Patients with an estimated glomerular filtration rate (eGFR) of less than 20 ml/min/1.73 m² or patients on dialysis.
* Chronic Anticoagulation Therapy: Patients requiring chronic oral anticoagulation (e.g., warfarin, DOACs) beyond DAPT.
* Thrombocytopenia: Platelet count less than 100,000/mm³.
* Contraindications to Antiplatelet Therapy: Allergy or intolerance to aspirin or P2Y12 inhibitors.
* Liver Disease: Patients with cirrhosis or significant liver dysfunction.
* Limited Life Expectancy: Patients with a life expectancy of less than 12 months due to other non-cardiac conditions.
* Other Medical Conditions: Any condition that might interfere with adherence to the study protocol or follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3566 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Cardiovascular and Cerebrovascular Events (NACCE) within 12 Months Post-PCI | 12 months of enrollment
  NACCE is a composite of major adverse cardiovascular events (MACEs) and cerebrovascular events, and any significant bleeding event (classified according to BARC 2-5). Cumulative risk of NACCE will be compared between the 1-month DAPT and 12-month DAPT groups.

SECONDARY OUTCOMES:
12-month Target Vessel Failure (TVF) Rate | 12 months of enrollment
  TVF is defined as a composite of target vessel myocardial infarction (TVMI), target vessel revascularization (TVR), or cardiovascular death related to the target vessel. Cumulative incidence of TVF will be compared between each treatment group.
12-month Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 12 months of enrollment
  MACCE includes cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and clinically-driven revascularization or definite stent thrombosis.
  Cumulative risk of MACCE will be compared between the 1-month DAPT and 12-month DAPT groups.
Major Bleeding Events Classified by BARC (Bleeding Academic Research Consortium) Scale | 12 months of enrollment
  To compare the rate of significant bleeding, classified according to the Bleeding Academic Research Consortium (BARC) types 2 to 5, between the two groups.
Clinical Characteristics of PCI Patients at Baseline (Descriptive Analysis of Demographics and Clinical Data) | 12 months of enrollment
  This outcome measure will include a detailed analysis of the clinical characteristics of patients undergoing PCI. The data will include demographics (age, gender), cardiovascular risk factors (diabetes, hypertension, smoking status), previous cardiovascular events, and other relevant clinical history such as comorbidities. Data will be summarized as means (for continuous variables like age) or percentages (for categorical variables like gender and risk factors). This measure aims to provide a baseline comparison between the two study groups (1-month DAPT vs. 12-month DAPT)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No